CLINICAL TRIAL: NCT02851277
Title: A Phase 1, Randomized, Placebo Controlled Study to Evaluate Safety, Tolerability and Immune Response in Adults Allergic to Peanut After Receiving Intradermal or Intramuscular Administration of ASP0892 (ARA LAMP Vax), a Single Multivalent Peanut (Ara h1, h2, h3) Lysosomal Associated Membrane Protein DNA Plasmid Vaccine
Brief Title: A Study to Evaluate Safety, Tolerability and Immune Response in Adults Allergic to Peanut After Receiving Intradermal or Intramuscular Administration of ASP0892 (ARA-LAMP-vax), a Single Multivalent Peanut (Ara h1, h2, h3) Lysosomal Associated Membrane Protein DNA Plasmid Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0892-CL-1001
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Peanut Allergy
Keywords: Peanut Allergy; ASP0892
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Low dose ASP0892 Intradermal (Experimental): Participants will receive study drug once every 2 weeks for a total of 4 doses. After participants complete the Low dose arms, the Dose Escalation Committee (DEC) will determine if the study can progress to the parallel higher dose arms.
  Interventions: Drug: ASP0892 Intradermal
- High dose ASP0892 Intradermal (Experimental): Participants will receive study drug once every 2 weeks for a total of 4 doses.
  Interventions: Drug: ASP0892 Intradermal
- Placebo Intradermal (Placebo Comparator): Participants will receive comparable Placebo once every 2 weeks for a total of 4 doses.
  Interventions: Drug: Placebo Intradermal
- High dose ASP0892 Intramuscular (Experimental): Participants will receive study drug once every 2 weeks for a total of 4 doses.
  Interventions: Drug: ASP0892 Intramuscular
- Placebo Intramuscular (Placebo Comparator): Participants will receive comparable Placebo once every 2 weeks for a total of 4 doses.
  Interventions: Drug: Placebo Intramuscular

INTERVENTIONS:
Drug: ASP0892 Intradermal — Intradermal injection
  Arms: High dose ASP0892 Intradermal; Low dose ASP0892 Intradermal
Drug: ASP0892 Intramuscular — Intramuscular injection
  Arms: High dose ASP0892 Intramuscular
Drug: Placebo Intradermal — Intradermal injection
  Arms: Placebo Intradermal
Drug: Placebo Intramuscular — Intramuscular injection
  Arms: Placebo Intramuscular

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ASP0892 after intradermal or intramuscular injection in adults with peanut allergy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) ≥ 18 and 32 at screening.
* Subject has a physician-diagnosed peanut allergy or history of peanut allergy. Subjects with history of nonsevere anaphylaxis (Grade ≤ 3) to peanuts (including mild wheezing or dyspnea without hypoxia) will be enrolled.
* Subject has an anti-Ara h2 IgE measured by ImmunoCAP > 0.35 kU/L.
* Subject has a positive SPT to peanut with a change in wheal diameter ≥ 3 mm as compared to a negative control.
* Subject has a positive peanut double-blinded placebo-controlled food challenge (DBPCFC) at Screen 2 visit with an eliciting dose ≤ 300 mg peanut protein (≤ 444 mg cumulative reactive dose [CRD]).
* Female subject must either:

  * Be of non-child bearing potential: post-menopausal (defined as at least 1 year without any menses) prior to screening, or documented surgically sterile.
  * Or, if of childbearing potential: Agree not to become pregnant during the study; and have a negative (urine) pregnancy test result at screening and at day 1 (predose); and, if heterosexually active, agree to consistently use 2 forms of highly effective birth control (at least one of which must be a barrier method) starting at screening and throughout the study period.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Male subject and female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (at least one of which must be a barrier method) starting at screening and continue throughout the study period, and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period, and for 90 days after the final study drug administration.

Exclusion Criteria:

* Subject has severe anaphylaxis to peanuts (Grades 4 or 5 including dyspnea associated with hypoxia, cyanosis, hypotension, or neurological compromise) per the Grading of Food-Induced Anaphylaxis According to Severity of Clinical Symptoms based on historical clinical symptoms.
* Subject develops a Grade 4 or 5 reaction during the DBPCFC.
* Subject who has received or is planning to receive administration of any vaccine (other than injectable Influenza vaccine) within 28 days prior to the administration of the study vaccine or at any time during the study.
* Subject who received any specific immunotherapy for allergy (e.g., epicutaneous immunotherapy [EPIT], sublingual immunotherapy [SLIT], subcutaneous immunotherapy [SCIT], and oral immunotherapy [OIT]) during the past 12 months, currently, or plans to receive during the course of the study.
* Subject who has used the following drug(s) prior to the dosing of the study vaccine:

  * Within 2 months prior to study vaccine administration: Systemic (or inhaled) steroid, chemical mediator-isolation inhibitor, Th2 cytokine inhibitor, thromboxane A2 synthesis inhibitor, thromboxane A2 receptor antagonist, β-blocker, angiotensin-converting enzyme inhibitors, and/or angiotensin-receptor blockers
  * Within 3 months prior to study vaccine administration: Biologics and/or immune modulators (including anti-TNFα antibody and anti-IgE monoclonal antibody)
* Subject who has history of allergic reactions such as anaphylactic shock, angioedema with airway constriction or hypotension caused by food other than peanut and/or medical products (including vaccine) in the past.
* Subject's laboratory test results at screening or prior to study vaccine dosing on day 1 are outside the normal limits and considered to be clinically significant.
* Subject with anti-LAMP-1 antibodies above the cut-point for the Tier 1 assay and who is confirmed positive in the Tier 2 assay at Screen 1 visit (baseline).
* Subject who had a positive test results for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen/ antibody.
* Subject who has immune disorders (including autoimmune disease) and/or diseases requiring immunosuppressive drugs.
* Subject who was diagnosed with immunodeficiency in the past.
* Subject who has uncontrolled hypertension.
* Subject who has a history of cardiovascular disease, arrhythmias, chronic lung disease, active eosinophilic gastrointestinal disease, or any other medical or surgical conditions which places the subject at increased risk for participation in the study.
* Subject who has a complication or medical history of respiratory disease which requires medical treatment.
* Subject who has a complication or medical history of malignant tumor.
* Subject who has mental conditions such as schizophrenia, bipolar disorder, and major depressive disorder, or a subject who has received drug(s) for the treatment of dementia.
* Subject who has severe or poorly controlled dermatitis atopic or generalized eczema.
* Subject who is unable to discontinue antihistamines within 7 days or 5 half-lives (whichever duration is longer) as follows:

  * prior to dosing through 7 days post last dose of study vaccine
  * prior to skin prick testing and oral food challenge procedures
* Subject who has asthma other than mild intermittent asthma (National Heart, Lung, and Blood Institute [NHLBI] guidelines) and has a FEV1 value < 80% and/or requiring chronic maintenance treatment (i.e., inhaled corticosteroids).
* Subject who has already received vaccination of LAMP-vax such as ASP0892.
* Subject who has received investigational therapy within 35 days or 5 half- lives whichever is longer, prior to screening.
* Subject who is an employee of the Astellas Group or vendors involved in the study.
* Subject who has any condition which makes the subject unsuitable for study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by number of participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 360
Safety as assessed by Vital sign: body temperature | Up to Day 360
Safety as assessed by Vital sign: blood pressure | Up to Day 360
Safety as assessed by Vital sign: pulse rate | Up to Day 360
Safety as assessed by 12- lead Electrocardiograms (ECGs) | Up to Day 360
  The overall conclusion will be recorded as normal and abnormal (not clinically significant/ clinically significant).
Safety as assessed by Laboratory test: hematology | Up to Day 360
Safety as assessed by Laboratory test: biochemistry | Up to Day 360
Safety as assessed by Laboratory test: urinalysis | Up to Day 360
Safety as assessed by Anti-Lysosomal associated membrane protein-1 (LAMP-1) antibody | Up to Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (8):
- United States (8):
  - Site US10014, Little Rock, Arkansas
  - Site US10008, Mountain View, California
  - Site US10001, Baltimore, Maryland
  - Site US10002, Boston, Massachusetts
  - Site US10004, New York, New York
  - Site US10003, Chapel Hill, North Carolina
  - Site US10012, Cincinnati, Ohio
  - Site US10006, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Ferslew BC, Smulders R, Zhu T, Blauwet MB, Kusawake T, Spence A, Aldridge K, DeBerg HA, Khosa S, Wambre E, Chichili GR. Safety and immunopharmacology of ASP0892 in adults or adolescents with peanut allergy: two randomized trials. Allergy. 2024 Feb;79(2):456-470. doi: 10.1111/all.15931. Epub 2023 Nov 27. PMID 38010254
- [Derived] Reyes AJ, Hosein AS, Ramcharan K, Perot S. Anaphylaxis and other allergic reactions to food: a global challenge. BMJ Case Rep. 2020 May 14;13(5):e231425. doi: 10.1136/bcr-2019-231425. PMID 32414772
- See also: Link to results on the Astellas Clinical Study Results website. — https://www.clinicaltrials.astellas.com/study/?pid=0892-CL-1001